CLINICAL TRIAL: NCT06945887
Title: Treatment of Desmoid Fibromatosis With Arterial Embolization: Retrospective and Prospective Observational Study
Brief Title: Treatment of Desmoid Fibromatosis With Arterial Embolization
Acronym: TAE-DESMO
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CE AVEC: 49/Oss/IOR
Record Dates: First submitted 2025-04-18; First posted 2025-04-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Desmoid Fibromatosis
Keywords: Desmoid fibromatosis; Embolization
MeSH Terms: conditions — Desmoid Tumors | interventions — Embolization, Therapeutic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Performed embolization
  Interventions: Procedure: embolization therapy

INTERVENTIONS:
Procedure: embolization therapy — Identification of the main vessels afferent to the tumor to be treated. -Selective and super-selective catheterization of pathological arterial branches, responsible for the blood supply to the neoplasm, through the use of micro-catheters. - Injection of embolizing material (hydrogel microspheres) - Control of technical success: the embolization will be followed by diagnostic arteriography that will evaluate the success of the procedure (occlusion of more than 90 percent of the pathologic vasculature).

SUMMARY:
Desmoid fibromatoses are rare and locally aggressive mesenchymal tumors. The current scientific evidence regarding the efficacy and safety of the treatment of desmoid fibromatosis by arterial embolization is constituted by several retrospective and prospective studies. These studies report promising results through the use of chemoembolization, that is, arterial embolization using particles loaded with chemotherapy.

Instead, the type of treatment we propose would consist of injection of embolizing material without the use of chemotherapy, based on the positive results we have consistently reported over the years on arterial embolization of musculoskeletal tumors.

DETAILED DESCRIPTION:
Desmoid fibromatoses are rare (1-2 cases/million per year) and locally aggressive, characterized histologically by monoclonal myoblasts present in abundant stromal tissue.The current therapeutic strategy has abandoned primary resection, as recurrences after resection are common and often their phenotype is more infiltrative. Nonsurgical approaches remain suboptimal. For asymptomatic disease, current guidelines suggest an initial period of active surveillance. The current scientific evidence regarding the efficacy and safety of the treatment of desmoid fibromatosis by arterial embolization is constituted by several retrospective and prospective studies. These studies report promising results through the use of chemoembolization, that is, arterial embolization using particles loaded with chemotherapy.

Instead, the type of treatment we propose would consist of injection of embolizing material without the use of chemotherapy, based on the positive results we have consistently reported over the years on arterial embolization of musculoskeletal tumors.

Doxorubicin is routinely used in the treatment of soft tissue sarcomas and other mesenchymal malignancies. Its use against desmoid fibromatosis is effective but associated with hematologic, gastrointestinal, and cardiac toxicity. Consequently, this drug is reserved for symptomatic, nonresponsive, rapidly growing, or life-threatening fibromatoses.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged ≥ 12 years
* Fibromatosis demsoid symptomatic and in active phase (documented growth at last follow-ups)
* Patients not eligible for surgery or cryoablation
* Patients who have had embolization surgery for fibromatosis desmoide from 01/01/2023 to date and all new patients listed for this type of treatment.
* Signature of informed consent to the study

Exclusion Criteria:

* Patients with life expectancy <3 months or severely impaired status functional status (ASA 4)
* Patients with fibromatosis not in active phase, documented clinically and by investigations imaging (MRI, CT)
* Patients with coagulation deficiency or plateletopenic disease
* Patients with documented active infection
* Incompatibility to performing MRI examination.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by desmoid fibromatoses eligible to be treated with transarterial embolization
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain (VAS score) | 1 year
  Clinical assessment regarding pain by Visual Analogue Scale (VAS) score (0-100 mm), in which 0 represents no pain, and 100 represents maximum pain imaginable.
Reduction of antalgic therapy (mg) | 1 year
  Mean reduction in the use of pain medications evaluated in mg of active ingredient taken daily before the treatment and at follow-up.
Volume reduction in cm³ | 1 year
  Reduction of the lesion evaluated with MRI, measuring the diameter of the lesion in cm³.

SECONDARY OUTCOMES:
Improvement in quality of life (EORTC QLQ-C15-PAL questionnaire) | 1 year
  Clinical assessment regarding quality of life by EORTC QLQ-C15-PAL questionnaire. The questionnaire consists of several scales, covering different aspects related to palliation. The maximum and minimum scores for each scale of the questionnaire can range from 0 to 100. The interpretation of scores depends on the specific scale in the questionnaire, and a higher value may indicate either greater negative impact (e.g., more symptoms or more suffering) or greater positive impact (e.g., better quality of life or less symptomatology).
Improvement in quality of life (EORTC QLQ - BM22) | 1 year
  Clinical assessment regarding quality of life by EORTC QLQ - BM22 questionnaire. The questionnaire consists of several scales, covering different aspects related to palliation. The maximum and minimum scores for each scale of the questionnaire can range from 0 to 100. The interpretation of scores depends on the specific scale in the questionnaire, and a higher value may indicate either greater negative impact (e.g., more symptoms or more suffering) or greater positive impact (e.g., better quality of life or less symptomatology). The overall assessment requires a detailed analysis of individual scores and related scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No